CLINICAL TRIAL: NCT07180459
Title: The Treatment of Unresectable Liver Cancer With Graded Embolization of Uniform-sized Drug-loaded Microspheres Combined With Donafenib：A Prospective, Single-arm, Multicenter, Observational Study
Brief Title: The Treatment of Unresectable Liver Cancer With E-TACE Combined With Donafenib：A Prospective, Single-arm, Multicenter, Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Xuhua Duan (Other)
Responsible Party: Sponsor-Investigator, Xuhua Duan, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Other Study IDs: 2025-KY-1085-002
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma; Carcinoma, Hepatocellular | interventions — donafenib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- E-TACE in Combination with Donafenib
  Interventions: Procedure: E-TACE; Drug: Donafenib

INTERVENTIONS:
Procedure: E-TACE — The 70/100μm drug-loaded microspheres were loaded with anthracyclines (30mg-50mg Idarubicin) at 2mL, and then combined with non-isoionic contrast agents to embolize the tumor supplying arteries, and then 250μm or 400μm drug-loaded microspheres were loaded anthracyclines (30mg-50mg Idarubicin) with 2mL/3mLto embolize the tumor supplying arteries at different grades and diameters.
Drug: Donafenib — 400mg QD

SUMMARY:
To clarify the safety and efficacy of using uniform-sized drug-loaded embolic microspheres (E-TACE) of different particle sizes for graded embolization during TACE combined with Donafenib in the treatment of unresectable primary liver cancer. To determine whether this therapy can prolong the ORR, DCR, PFS, OS and other indicators.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with unresectable primary liver cancer who strictly meet the clinical diagnostic criteria of the "Primary Liver Cancer Diagnosis and Treatment Guidelines" (2024 Edition) or who have been diagnosed through pathological histology or cytology examination, and who have at least one measurable lesion (according to the mRECIST 1.1 version, the long diameter of the measurable lesion on spiral CT scan should be ≥ 10mm or the short diameter of the enlarged lymph node should be ≥ 15mm); (2) Tumor staging: CNLC stage Ib, IIa, IIb, IIIa, IIIb or BCLC A, B, C stage; non-diffuse liver cancer (PVTT classified according to the Japanese Liver Cancer Research Society's portal vein tumor thrombus characteristics as Vp1/2, Vp3, Vp4); (3) Gender of the patients is not restricted, and the age is 18-80 years old; expected lifespan is ≥ 3 months; (4) Within 1 week before enrollment, the ECOG PS score: 0-1; (5) No severe comorbidities, such as hypertension, coronary heart disease and history of mental illness, no severe allergy history; (6) Liver function should reach Child-Pugh grade A or B; (7) Laboratory tests meet the following requirements: platelets ≥ 50×109/L; hemoglobin ≥ 9g/dL; white blood cells ≥ 4×109/L; neutrophils ≥ 1.5×109/L); serum total bilirubin ≤ 1.5 times the upper limit of normal value (ULN), transaminases (ALT, AST) ≤ 5 times ULN; creatinine ≤ 1.5 times ULN; urine routine shows urine protein < 2+; for patients whose urine protein ≥ 2+ at baseline, 24-hour urine collection should be conducted and the 24-hour urine protein quantification < 1g; international normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN; (8) HBV DNA < 2000 IU/ml (104 copies/ml); (9) For pregnant women of childbearing age, a pregnancy test should be conducted within 7 days before enrollment; (10) Patients have signed the informed consent form agreeing to participate in this trial study; good compliance and cooperation with treatment.

Exclusion Criteria:

* (1) Imaging examination shows that the liver tumor is huge (≥ 60% of liver volume), or there is a main portal vein tumor thrombus (occupying the vascular diameter ≥ 50%), or the tumor thrombus invades the mesenteric vein or inferior vena cava, or there are obvious native hepatic artery - portal vein fistulas and native hepatic artery - hepatic vein fistulas that cannot safely use drug-loaded microspheres; (2) Before participating in this study, they have undergone local treatments such as traditional TACE, thermal ablation, cryoablation, external radiotherapy and radioactive particle implantation, and have received systemic chemotherapy, oral liver cancer targeted drugs (sorafenib, lenafolate, apatinib) and immune therapy (PD-1/PD-L1/CDLA-4/biologic double therapy); (3) Patients with diffuse liver cancer; known hepatocellular carcinoma and mixed cell carcinoma and fibroplastic cell carcinoma; having other untreated malignant tumors in the past (within 5 years) or simultaneously; except for cured skin basal cell carcinoma and cervical carcinoma in situ; (4) Having grade II or above myocardial ischemia or myocardial infarction, and uncontrolled arrhythmia (including QTc interval for males ≥ 450ms, females ≥ 470ms); (5) Having a history of gastrointestinal bleeding in the past 6 months or having a clear tendency for gastrointestinal bleeding, such as: esophageal varices with bleeding risk, local active ulcer lesion, fecal occult blood ≥ (++), not eligible for inclusion; if fecal occult blood (+), a gastroscopy examination is required; (6) Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds), bleeding tendency or undergoing thrombolysis or anticoagulation treatment; (7) Patients with central nervous system metastasis or known brain metastasis; having objective evidence of past and current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of pulmonary function; patients with combined HIV infection; pregnant or lactating patients; patients preparing for liver transplantation (except for patients who have undergone liver transplantation in the past); (8) Severe systemic failure, with an expected survival period < 3 months; (9) Severe renal dysfunction (creatinine > 2mg/dl or creatinine clearance rate < 30ml/min); (10) Unable to complete the treatment plan due to various reasons, and lost follow-up within three months after enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 118 Hepatocellular carcinoma Patients
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 1 year
  The definition of PFS is the time from the first administration of combined therapy to the first imaging assessment indicating tumor progression or death, whichever occurs first.

SECONDARY OUTCOMES:
ORR | up to 1 year
  ORR is defined as the proportion of patients who achieve complete remission (CR, Complete Response) and partial remission (PR, Partial Response) according to the mRECIST criteria
OS | up to1 year
  The OS is defined as the time from the first administration of combined therapy to the occurrence of any cause of death. If there is no death record for the patient, the last visit time will be used as the censored value.
TTP | up to1 year
  The TTP is defined as the time from the first administration of combined therapy to the first imaging assessment revealing tumor progression
AE | up to1 year
  Adverse Events

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - People's Hospital of Kaiyang County, Guiyang, Guizhou
  - The Second Affiliated Hospital of Hainan Medical Universsity, Haikou, Hainan
  - Huai He Hospital of Henan University, Kaifeng, Henan
  - Luo He Central Hospital, Luohe, Henan
  - Luo Yang Central Hospital, Luoyang, Henan
  - Deng zhou People's Hospital, Nanyang, Henan
  - First People's Hospital of Shangqiu, Shangqiu, Henan
  - Zhou Kou Central Hospital, Zhoukou, Henan
  - Jiangxi Provincial People's Hospitail, Nanchang, Jiangxi
  - Second People's Hospital of Jiaozuo, Jiaozuo